CLINICAL TRIAL: NCT00222612
Title: Medical Research Council Working Party on Leukaemia in Children UK National Acute Lymphoblastic Leukaemia (ALL) Trial: UKALL 2003
Brief Title: Medical Research Council (MRC) Working Party on Leukaemia in Children UK National Acute Lymphoblastic Leukaemia (ALL) Trial: UKALL 2003
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Dr Vora, Sheffield University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKALL2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A or B with 2DI (Active Comparator): 3 or 4 drug induction plus 2 delayed intensifications
  Interventions: Drug: Standard childhood UK ALL protocol
- C plus 2DI (Experimental): Intensified treatment including Capizzi maintenance
  Interventions: Drug: Intensified treatment including Capizzi maintenance
- A or B with 1DI (Experimental): Reduced intensity treatment
  Interventions: Other: Reduced intensification

INTERVENTIONS:
Other: Reduced intensification — Deletion of one 7 week treatment block containing dexamethasone, vincristine, doxorubicin, Peg-asparaginase, intrathecal methotrexate, cyclophosphamide, cytarabine.
  Other Names: Removal of second delayed intensification
  Arms: A or B with 1DI
Drug: Standard childhood UK ALL protocol — No additional treatment to standard protocol.
  Arms: A or B with 2DI
Drug: Intensified treatment including Capizzi maintenance — Augmented consolidation: vincristine, Peg-asparaginase. Capizzi maintenance: iv methotrexate and peg-asparaginase
  Arms: C plus 2DI

SUMMARY:
A randomised trial for children with acute lymphoblastic leukemia, using the detection of minimal residual disease to define risk groups, aiming to answer the questions:

1. Can treatment be reduced without compromising efficacy in a MRD-defined low risk group?
2. Does further post-remission intensification improve outcome for a MRD-defined high risk group?
3. Measure the Quality of Life impact of the different treatment arms on the children and their families.

DETAILED DESCRIPTION:
Randomisations

Patients will be assigned to MRD risk groups based on day 29 and post consolidation MRD results and randomised as follows:

1. MRD Low Risk Group (MRD negative at day 29 and week 11 or positive <1 x 10-4 at day 28 and negative at week 11) will continue on previously assigned Regimens (A or B) but randomised between two delayed intensifications and one delayed intensification.
2. MRD High Risk Group (MRD positive > 1 x 10-4 at day 29) randomised between previously assigned Regimen (A or B) and Regimen C.
3. MRD Indeterminate Group (No MRD result or MRD positive <1 x 10-4 at day 29 and at week 11) will continue on previously assigned Regimen (A or B) and received two delayed intensifications

ELIGIBILITY:
Inclusion criteria:

Children aged 1 - 18 years with ALL except the following:

Exclusion criteria:

1. Infants less than a year old should be entered onto the Interfant ALL study.
2. Children with B-ALL (Burkitt-like, t(8;14), L3 morphology, SMIg positive). Patients with this disease will be eligible for the current UKCCSG B cell NHL/ALL trial.
3. Children with Philadelphia-positive ALL (t(9;22) or BCR/ABL positive) will start induction therapy on this protocol but transfer to the European Intergroup Protocol as soon as their Philadelphia status is known.

Initially, eligible patients will be stratified into three risk groups based on the following criteria:

1. Standard risk: all children >1<10 years with a highest white cell count before starting treatment of <50x109/l, and who do not have BCR-ABL, hypodiploidy (≥44 chromosomes), or an MLL gene rearrangement.
2. Intermediate risk: all children ≥10 years old, or with a diagnostic WBC ≥50x109/l (or both) and who do not have BCR-ABL, hypodiploidy (≥44 chromosomes), or an MLL gene rearrangement.
3. High Risk: all children, irrespective of initial risk category, who have a slow early response (SER) as defined below - see section 6 - together with those who have BCR-ABL (induction only), hypodiploidy (≥44 chromosomes), or an MLL gene rearrangement. These patients will not be eligible for MRD randomisation.

Patients will then start treatment according to their risk group as follows:

1. Standard risk, (around 60-65% of the total): regimen A - three-drug induction.
2. Intermediate risk, (around 20- 30% of the total): regimen B - four-drug induction.
3. High risk (around 10-12% of the total): These patients will not be eligible for MRD randomisation. They will be allocated regimen C - four drug induction, augmented BFM consolidation, Capizzi interim maintenance, and two further BFM-style intensification periods of extended duration.

Inclusion criteria for entry into the randomisations:

1. Standard or Intermediate Risk as defined above.
2. Morphological Complete Remission (BM1 Marrow) at Day 29 of Induction.
3. Availability of MRD results at Day 28 and after consolidation therapy.
4. Informed consent obtained.
5. Induction given as protocol.

Exclusion criteria for entry into the MRD randomisation:

1. High Risk as defined above. These patients will receive Regimen C.
2. Day 28 non-remitters. These patients will receive Regimen C if BM2 or go off-protocol if BM3 (see below for definitions of BM2 and BM3).
3. MRD Indeterminate Group (No result or MRD positive < 1 x 10-4 at day 28 and after consolidation therapy) will continue on previously assigned therapy.
4. Sub-optimal induction therapy. The clinical significance of day 28 MRD is uncertain in patients who have received sub-optimal induction therapy. Please discuss these patients with a co-ordinator.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2100 (Estimated)
Dates: Start 2003-10; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 5 years

SECONDARY OUTCOMES:
Survival | 5 years
Quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Vora, Principal Investigator — Sheffield Children's Hospital
Locations (1):
- Sheffield Children's Hospital, Sheffield, United Kingdom

REFERENCES:
- [Derived] Moorman AV, Antony G, Wade R, Butler ER, Enshaei A, Harrison CJ, Moppett J, Hough R, Rowntree C, Hancock J, Goulden N, Samarasinghe S, Vora A. Time to Cure for Childhood and Young Adult Acute Lymphoblastic Leukemia Is Independent of Early Risk Factors: Long-Term Follow-Up of the UKALL2003 Trial. J Clin Oncol. 2022 Dec 20;40(36):4228-4239. doi: 10.1200/JCO.22.00245. Epub 2022 Jun 17. PMID 35714315
- [Derived] Wilson K, Case M, Minto L, Bailey S, Bown N, Jesson J, Lawson S, Vormoor J, Irving J. Flow minimal residual disease monitoring of candidate leukemic stem cells defined by the immunophenotype, CD34+CD38lowCD19+ in B-lineage childhood acute lymphoblastic leukemia. Haematologica. 2010 Apr;95(4):679-83. doi: 10.3324/haematol.2009.011726. Epub 2009 Nov 30. PMID 19951974
- See also: Related Info — http://www.ctsu.ox.ac.uk